CLINICAL TRIAL: NCT06575595
Title: A Pharmacokinetic Study of Tulisokibart Administered Subcutaneously Via Autoinjector or Syringe in Healthy Adult Participants
Brief Title: Pharmacokinetic (PK) Characterization of Subcutaneous Tulisokibart (MK-7240-010)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7240-010; MK-7240-010 (Other: MSD)
Record Dates: First submitted 2024-08-16; First posted 2024-08-28 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Single dose delivered subcutaneously (SC) with an autoinjector
  Interventions: Biological: Tulisokibart
- Treatment B (Experimental): Single dose of concentration A delivered SC with syringe and vial
  Interventions: Biological: Tulisokibart
- Treatment C (Experimental): Single dose of concentration B delivered SC with syringe and vial
  Interventions: Biological: Tulisokibart

INTERVENTIONS:
Biological: Tulisokibart — single dose via SC autoinjector (Treatment A) or concentration A or concentration B SC injection via syringe and vial (Treatments B and C)
  Other Names: MK-7240

SUMMARY:
The primary objectives of the study are to characterize the pharmacokinetics (PK) of a single subcutaneous (SC) dose of tulisokibart (MK-7240) administered via autoinjector (AI) (Treatment A) and to characterize the PK of different concentrations of tulisokibart following SC administration of a single dose via vial/syringe (Treatments B and C). There is no formal hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Is in good health
* Has a body mass index (BMI) between 18 and 32 kg/m2, inclusive
* Has a weight between 50 and 100 kg, inclusive

Exclusion Criteria:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of clinically significant psychiatric disorder of the last 5 years
* Has a history of cancer (except fully treated non-melanoma skin cell cancers or cervical carcinoma in situ after complete surgical removal) within the last 5 years or has had diagnostic evaluation suggestive of malignancy (eg, chest or breast imaging) in which the possibility of malignancy cannot be reasonably excluded following additional clinical assessments
* Has a history of significant multiple and/or severe allergies (eg, food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (ie, systemic allergic reaction) to prescription or nonprescription drugs or food
* Has a positive test(s) for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or human immunodeficiency virus (HIV); OR positive hepatitis B core antibody (HBcAb) with negative hepatitis B core antibody (HBsAb)
* Has a history of more than one episode of herpes zoster infection or history of disseminated herpes zoster infection
* Has a history of or current active tuberculosis (TB) infection; history of latent TB that was not fully treated or a positive QuantiFERON-TB test at screening
* Is a smoker and/or has used nicotine or nicotine-containing products (eg, nicotine patch and electronic cigarette) within 3 months of screening
* Consumes greater than 3 servings of alcoholic beverages per day
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 12 months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve from Time 0 to Infinity (AUC0-inf): Treatment A | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the AUC0-inf of tulisokibart. AUC0-inf is defined as the area under concentration-time curve of tulisokibart from time zero to infinity.
Area Under the Curve from Time 0 to Last Measurable Concentration (AUC0- last): Treatment A | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the AUC0-last of tulisokibart. AUC0-last is defined as the area under the concentration-time curve from time zero to time of last measurable concentration of tulisokibart.
Maximum Plasma Concentration (Cmax): Treatment A | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the Cmax of tulisokibart. Cmax is defined as the maximum concentration of tulisokibart reached.
Time to Cmax (Tmax): Treatment A | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the Tmax of tulisokibart. Tmax is defined as the time to maximum concentration of tulisokibart reached.
Clearance after Nonintravenous Administration (CL/F): Treatment A | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the CL/V of tulisokibart. CL/F is the rate at which the tulisokibart is completely removed from plasma.
Volume of Distribution (V/F): Treatment A | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the V/F of tulisokibart. V/F is the volume of distribution of tulisokibart.
Half Life (t1/2): Treatment A | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the t1/2 of tulisokibart. t1/2 is defined as the time required to divide plasma concentration of tulisokibart by half.

SECONDARY OUTCOMES:
AUC0-inf: Treatment B vs Treatment C | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the AUC0-inf of tulisokibart. AUC0-inf is defined as the area under concentration-time curve of tulisokibart from time zero to infinity.
AUC0-last: Treatment B vs Treatment C | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the AUC0-last of tulisokibart. AUC0-last is defined as the area under the concentration-time curve from time zero to time of last measurable concentration of tulisokibart.
Cmax: Treatment B vs Treatment C | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the Cmax of tulisokibart. Cmax is defined as the maximum concentration of tulisokibart reached.
Tmax: Treatment B vs Treatment C | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the Tmax of tulisokibart. Tmax is defined as the time to maximum concentration of tulisokibart reached.
CL/V: Treatment B vs Treatment C | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the CL/V of tulisokibart. CL/F is the rate at which the tulisokibart is completely removed from plasma.
V/F: Treatment B vs Treatment C | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the V/F of tulisokibart. V/F is the volume of distribution of tulisokibart.
t1/2: Treatment B vs Treatment C | Predose and Days 1, 2, 3, 4 ,5 ,6, 8, 10, 15, 29, 57, 71 and Post-study (Day 99)
  Blood will be collected at pre-specified time points to determine the t1/2 of tulisokibart. t1/2 is defined as the time required to divide plasma concentration of tulisokibart by half.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- QPS Missouri ( Site 0003), Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com